CLINICAL TRIAL: NCT04145830
Title: Efficacy and Safety of UCP in the Treatment of Primary Glaucoma in China
Brief Title: UCP Glaucoma Treatment for Primary Glaucoma in China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EyeTechCare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS18-CHN-04
Record Dates: First submitted 2019-10-29; First posted 2019-10-31 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2019-10

CONDITIONS: Glaucoma Treatment Using Focused Ultrasound
Keywords: Glaucoma, ciliary body, ultrasound
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ultrasound Cyclo Plasty (UCP) (Experimental): Ultrasound Cyclo Plasty (UCP) using focused ultrasound
  Interventions: Device: Ultrasound Cyclo Plasty (UCP)

INTERVENTIONS:
Device: Ultrasound Cyclo Plasty (UCP) — Cyclocoagulation using High Intensity Focused Ultrasound
  Other Names: UCP by EyeOP1 device

SUMMARY:
To collect safety and efficacy data on Ultrasound Cycle Plasty treatment (UCP) in primary glaucoma asian patients.

ELIGIBILITY:
Inclusion Criteria:

* Primary Open Angle and primary Angle Closure glaucoma
* Subject where the IOP is not adequately controlled with glaucoma medication, and can not or not agree for incisional glaucoma surgery
* IOP ≥ 21 mmHg and ≤ 40 mmHg
* Best Corrected Visual Acuity > Hand Motion
* Patient able and willing to sign the informed consent and complete postoperative followup requirements

Exclusion Criteria:

* History of ocular or retrobulbar tumor
* Ocular infection within 14 days prior to the procedure of Ultrasound Cyclo Plasty (UCP)
* History of Cyclo-destructive procedures (cryotherapy, Laser transscleral cyclophotocoagulation; Laser endophotocoagulation)
* Congenital glaucoma
* History of ciliary body surgery or vitrectomy in the study eye
* Ocular disease other than glaucoma that may affect assessment of visual acuity and/or IOP (choroidal hemorrhage or detachment, lens subluxation, thyroid ophthalmopathy, proliferative diabetic retinopathy, clinical significant macular edema, retinal detachment)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-04-29 (Actual); Study Completion 2020-11-02 (Actual)

PRIMARY OUTCOMES:
Efficacy endpoint : reduction of the intraocular pressure | 6 months
  Reduction of the intraocular pressure relative to the preoperative value at each follow-up visits in mmHg and in % of reduction

SECONDARY OUTCOMES:
Safety endpoint: rate of per operative complications | 6 months
  Rate of per-operative device and/or procedure related adverse events
Safety endpoint: rate of post-operative complications | 6 months
  Rate of post-operative complications during the follow-up period
Efficacy endpoint: Number of ocular hypotensive medications | 6 months
  Mean number of IOP lowering medications at each visit during the follow-up period

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Shanghai Eye Diseases Prevention and Treatment Center - Department of Ophthalmology, Shanghai
  - E&ENT Fudan University, Shanghai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aptel F, Denis P, Rouland JF, Renard JP, Bron A. Multicenter clinical trial of high-intensity focused ultrasound treatment in glaucoma patients without previous filtering surgery. Acta Ophthalmol. 2016 Aug;94(5):e268-77. doi: 10.1111/aos.12913. Epub 2015 Nov 7. PMID 26547890
- [Background] Torky MA, Al Zafiri YA, Hagras SM, Khattab AM, Bassiouny RM, Mokbel TH. Safety and efficacy of ultrasound ciliary plasty as a primary intervention in glaucoma patients. Int J Ophthalmol. 2019 Apr 18;12(4):597-602. doi: 10.18240/ijo.2019.04.12. eCollection 2019. PMID 31024813
- [Background] De Gregorio A, Pedrotti E, Stevan G, Montali M, Morselli S. Safety and efficacy of multiple cyclocoagulation of ciliary bodies by high-intensity focused ultrasound in patients with glaucoma. Graefes Arch Clin Exp Ophthalmol. 2017 Dec;255(12):2429-2435. doi: 10.1007/s00417-017-3817-4. Epub 2017 Oct 17. PMID 29043438
- [Background] Posarelli C, Covello G, Bendinelli A, Fogagnolo P, Nardi M, Figus M. High-intensity focused ultrasound procedure: The rise of a new noninvasive glaucoma procedure and its possible future applications. Surv Ophthalmol. 2019 Nov-Dec;64(6):826-834. doi: 10.1016/j.survophthal.2019.05.001. Epub 2019 May 22. PMID 31125570
- [Background] Giannaccare G, Vagge A, Sebastiani S, Urbini LE, Corazza P, Pellegrini M, Carmassi L, Bergamini F, Traverso CE, Campos EC. Ultrasound Cyclo-Plasty in Patients with Glaucoma: 1-Year Results from a Multicentre Prospective Study. Ophthalmic Res. 2019;61(3):137-142. doi: 10.1159/000487953. Epub 2018 May 16. PMID 29768281
- [Background] Pellegrini M, Sebastiani S, Giannaccare G, Campos EC. Intraocular inflammation after Ultrasound Cyclo Plasty for the treatment of glaucoma. Int J Ophthalmol. 2019 Feb 18;12(2):338-341. doi: 10.18240/ijo.2019.02.23. eCollection 2019. PMID 30809493
- [Background] Melamed S, Goldenfeld M, Cotlear D, Skaat A, Moroz I. High-intensity focused ultrasound treatment in refractory glaucoma patients: results at 1 year of prospective clinical study. Eur J Ophthalmol. 2015 Nov-Dec;25(6):483-9. doi: 10.5301/ejo.5000620. Epub 2015 May 13. PMID 25982212